CLINICAL TRIAL: NCT01628198
Title: Impact of Renal SympAthetic DenerVation on Chronic HypErtension
Acronym: SAVE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recommendation by the study's DSMB due to insufficient data to determine efficacy.
Sponsor: Vivek Reddy (Other)
Responsible Party: Sponsor-Investigator, Vivek Reddy, Director Cardiac Arrhythmia Service, Professor Of Medicine, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 12-0740
Record Dates: First submitted 2012-06-12; First posted 2012-06-26 (Estimated); Results first posted 2018-01-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Uncontrolled Hypertension
Keywords: Hypertension; renal denervation; renal ablation; uncontrolled high blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Renal denervation group (Experimental): Celcius Thermacool Catheter or Chilli II Cooled Ablation Catheter
  Interventions: Device: Celcius Thermacool Catheter or Chilli II Cooled Ablation Catheter

INTERVENTIONS:
Device: Celcius Thermacool Catheter or Chilli II Cooled Ablation Catheter — Saline-Irrigated Radiofrequency Ablation Catheter will be placed in the renal arteries in a circumferential manner and energy will be delivered to create 4 burn lesions.
  There are 2 devices that can be used---this is optional, based on physician preference:
  Celcius Thermacool Catheter Biosense Webster, Inc Diamond Bar, California
  or
  Chilli II Cooled Ablation Catheter Boston Scientific Corporation San Jose, California
  Other Names: Renal Ablation; Renal denervation

SUMMARY:
Despite the development of many drug therapies designed to treat high blood pressure (hypertension), it remains a considerable and poorly managed health, social and economic burden. For various reasons, including the high health care costs of treatment, there are estimates that up to 65% of patients with high blood pressure have untreated and/or uncontrolled blood pressure (BP).

Aside from its effect on kidney function, chronic high blood pressure increases the risk for stroke, and heart disease. It is also thought to be involved in the formation of irregular heartbeats. This link between high blood pressure and heart health has been well described, as has their combined effect on the aging and the obesity-battling Western world.

A recently published study (Symplicity HTN-2 trial) established the benefit of a new treatment procedure, catheter-based renal sympathetic denervation (RSDN) for hypertension, as having enormous potential for the treatment of patients with high blood pressure. This multi-center trial will attempt to confirm and expand on these promising data. Patients who enroll in the trial will be followed for 4 years.

DETAILED DESCRIPTION:
Aside from its obvious impact on renal function, chronic hypertension significantly increases the risk for stroke, coronary artery disease, heart failure, and vascular disease, and it is believed to mediate the pathogenesis and progression of cardiac arrhythmias via its remodeling effects on cardiac anatomy. This inextricable link between hypertension and cardiovascular health has been well described, as has their combined effect on up to 40% of the aging, obesity-battling Western world.

Despite the development of numerous anti-hypertensive drug therapies-diuretics, angiotensin-converting enzyme inhibitors, alpha-adrenergic blockers, angiotensin-receptor blockers, calcium-channel blockers, beta blockers, and vasodilators-designed to block various and multiple avenues of the complex renal-cardiovascular circuit, hypertension remains a considerable, and poorly managed, social and economic burden. For various reasons, including the enormous health care costs of treatment, up to 65% of hypertensive patients have untreated and/or uncontrolled blood pressure (BP). Of those with uncontrolled blood pressure, ~10% have resistant hypertension-defined as elevated BP refractory to treatment with 3 antihypertensive agents of different classes.

But an even greater problem than the ineffectiveness of available therapies is their applicability. As has been observed with other illnesses, patients are often the greatest obstacles to their own care. Convincing patients to adhere to a life-long regimen of expensive medication for something which causes no immediate, palpable impact to their lives, is a challenging feat for today's pressed-for-time physician.

Therefore, of particular interest and profound promise is a recent study examining the effects on chronic blood pressure management of catheter-based renal sympathetic denervation (Symplicity HTN-1, Krum et al, Lancet 373:1275, 2009). This proof-of-principle study revealed that the procedure could be performed safely and without any procedure-related sequelae in 50 patients with baseline office blood pressure of 177±20 / 101±15, on 4.7 anti-hypertensive medications. At 12 months post-procedure, the mean reduction in office blood pressures was a remarkable -27/-17 mm Hg, with a concurrent 47% reduction in renal noradrenaline spillover. Importantly, these favorable blood pressure results were maintained over 2 years (see Fig).

Then, Esler et al performed a multicenter, randomized controlled trial comparing catheter based renal denervation to optimal medication therapy in patients with drug-resistant hypertension (Symplicity HTN-2, Lancet 2010; 376:1903-1909). In this study of 106 randomized patients, the 6-month office BPs in the denervation group decreased by 32/12 mmHg (SD 23/11, baseline of 178/96 mmHg, p<0.0001), whereas they did not differ from baseline in the control group (change of 1/0 mmHg [SD 21/10], baseline 178/97 mmHg, p=N.S.). There were no serious procedure-related or device-related complications. And most recently, besides the hydrostatic effect on blood pressure, it was recently demonstrated that RSDN significantly reduces LV mass and improves diastolic function in patients with refractory hypertension (J Am Coll Cardiol 2012; 59:901-9). Together, these favorable effects all suggest that there may important beneficial prognostic implications for RSDN in patients with resistant hypertension at high cardiovascular risk.

But of note, in both Lancet studies, the catheter used for the renal ablation procedure was a specialized radiofrequency ablation catheter that is not yet FDA-approved. To this end, it has been demonstrated that RSDN can be safely performed in patients using an off-the-shelf solid-tip radiofrequency ablation catheter typically used for cardiac ablation (EuroIntervention 2012; 7(9):1077-80). In addition, we have recently demonstrated that a standard off-the-shelf irrigated radiofrequency ablation catheters can also be used to achieve a similar effect (H.Ahmed / P.Neuzil / V.Reddy, JACC-Cardiovasc Interven, in press). Briefly, in drug-refractory hypertension patients, an irrigated radiofrequency ablation catheter (Celsius Thermocool catheter, Biosense-Webster Inc, Diamond Bar, California) was used to perform bilateral renal arterial sympathetic denervation. Briefly, over a 6 month period, 1) the systolic/diastolic BPs (as determined by 24-hour blood pressure monitoring) decreased by -21/-11 mmHg (for comparison, the change in the 24-hour blood pressure change in Symplicity HTN-2 was -11/-7 mm Hg); 2) all patients experienced a decrease in systolic BP of at least 10 mm Hg (range: 10-40 mm Hg); 3) there was no evidence of renal artery stenosis or aneurysm at repeat angiography; and 4) there was a significant decrease in renal sympathetic activity at 3 months: including metanephrine (-12±4, p=0.003), normetanephrine (-18±4, p=0.0008) levels, and aldosterone levels (-60±33 ng/l, p=0.02). There was also no evidence of worsening renal function (change in serum creatinine was -1 mmol/L, p=0.4). These data provide the proof-of-principle that RSDN can be performed using an off-the-shelf saline-irrigated radiofrequency ablation catheter. [Of note, there were two major reasons that this off-the-shelf catheter was used: i) the lack of availability of the specialized RF ablation catheter used in the Lancet studies, and ii) unlike this specialized RF catheter, the catheter we employed had a saline-irrigated ablation element. In theory, saline-irrigation has the advantage of being less likely to cause thrombus or char formation during catheter ablation, and is also more likely to cause tissue surface sparing while ablating deeper tissue.] The purpose of this trial will be to evaluate the long term safety and efficacy of catheter-based renal sympathetic denervation in 500 hypertensive patients by following them for 2 years.

Study Rationale The recently published results of the Symplicity HTN-2 trial (Renal sympathetic denervation in patients with treatment resistant hypertension) establishing the therapeutic benefit of catheter-based renal sympathetic denervation for hypertension, have enormous potential for the management of a large and challenging patient population. The proposed prospective non-randomized multi-center trial will attempt to confirm and expand on these promising data by evaluating the long-term efficacy (and safety) of renal sympathetic denervation in patients with chronic hypertension. Patients who enroll in the trial will be followed for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 85 years of age.
* Refractory hypertension (per JNC-7, this is defined as BP ≥ 140/90 mmHg despite treatment with at least 3 anti-hypertensive drugs, at least one of which is a diuretic, or treatment by ≥ 4 anti-hypertensive drugs)
* Stable anti-hypertensive drug regimen, where no modifications have occurred for at least 2 weeks.
* Accessibility of renal vasculature.
* Ability to understand the requirements of the study.
* Willingness to adhere to study restrictions and comply with all post-procedural follow-up requirements.

Exclusion Criteria:

* Subject has a known secondary cause of hypertension.
* Subject has isolated White coat hypertension.
* Subject has Type 1 Diabetes.
* Subject has known significant renovascular abnormalities (e.g., significant renal artery stenosis, previous renal artery stenting or angioplasty that precludes the RSDN procedure because of no sites for ablation treatment, or the presence of an accessory renal artery in which the main renal artery is estimated to supply <75% of the kidney )
* Significant renal artery stenosis is defined as > 50% diameter stenosis on renal angiography. Per the guidelines for noninvasive vascular laboratory testing: a report from the American Society of Echocardiography and the Society for Vascular Medicine and Biology, significant renal artery stenosis is defined by any one of the following criteria on renal duplex ultrasound; i) Renal artery to aorta peak systolic velocity ratio ≥ 3.5; ii) Peak Systolic Velocity > 200 cm/s with evidence of post-stenotic turbulence; iii) end diastolic velocity >150 cm/s ; iv) Resistive Index (RI) > 0.8; v) An occluded renal artery demonstrates no flow in the affected vessel.
* Subject has hemodynamically significant valvular heart disease for which reduction of blood pressure would be considered hazardous.
* Subject has New York Heart Association (NYHA) Class III or IV congestive heart failure, due to either systolic or diastolic dysfunction.
* Subject has an eGFR<45 ml/min/1.73m2 (calculated by using the modified diet in renal disease (MDRD) formula), and is not receiving dialysis.
* Subject has orthostatic hypotension. (per the American Academy of Neurology/American Autonomic Society Conesus Statement, this is defined as a sustained reduction of systolic blood pressure of at least 20 mm Hg or diastolic blood pressure of 10 mm Hg within 3 min of standing or head-up tilt to at least 60° on a tilt table)
* Subject has a life expectancy < 1 year for any medical condition.
* Subject is currently enrolled in another investigational drug or device trial that would interfere with this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krum H, Schlaich M, Whitbourn R, Sobotka PA, Sadowski J, Bartus K, Kapelak B, Walton A, Sievert H, Thambar S, Abraham WT, Esler M. Catheter-based renal sympathetic denervation for resistant hypertension: a multicentre safety and proof-of-principle cohort study. Lancet. 2009 Apr 11;373(9671):1275-81. doi: 10.1016/S0140-6736(09)60566-3. Epub 2009 Mar 28. PMID 19332353
- [Background] Symplicity HTN-2 Investigators; Esler MD, Krum H, Sobotka PA, Schlaich MP, Schmieder RE, Bohm M. Renal sympathetic denervation in patients with treatment-resistant hypertension (The Symplicity HTN-2 Trial): a randomised controlled trial. Lancet. 2010 Dec 4;376(9756):1903-9. doi: 10.1016/S0140-6736(10)62039-9. Epub 2010 Nov 17. PMID 21093036
- [Background] Lloyd-Jones D, Adams R, Carnethon M, De Simone G, Ferguson TB, Flegal K, Ford E, Furie K, Go A, Greenlund K, Haase N, Hailpern S, Ho M, Howard V, Kissela B, Kittner S, Lackland D, Lisabeth L, Marelli A, McDermott M, Meigs J, Mozaffarian D, Nichol G, O'Donnell C, Roger V, Rosamond W, Sacco R, Sorlie P, Stafford R, Steinberger J, Thom T, Wasserthiel-Smoller S, Wong N, Wylie-Rosett J, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2009 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2009 Jan 27;119(3):480-6. doi: 10.1161/CIRCULATIONAHA.108.191259. No abstract available. PMID 19171871
- [Background] Kearney PM, Whelton M, Reynolds K, Muntner P, Whelton PK, He J. Global burden of hypertension: analysis of worldwide data. Lancet. 2005 Jan 15-21;365(9455):217-23. doi: 10.1016/S0140-6736(05)17741-1. PMID 15652604
- [Background] Sarafidis PA, Bakris GL. Resistant hypertension: an overview of evaluation and treatment. J Am Coll Cardiol. 2008 Nov 25;52(22):1749-57. doi: 10.1016/j.jacc.2008.08.036. PMID 19022154
- [Background] Cutler JA, Sorlie PD, Wolz M, Thom T, Fields LE, Roccella EJ. Trends in hypertension prevalence, awareness, treatment, and control rates in United States adults between 1988-1994 and 1999-2004. Hypertension. 2008 Nov;52(5):818-27. doi: 10.1161/HYPERTENSIONAHA.108.113357. Epub 2008 Oct 13. PMID 18852389
- [Background] Calhoun DA, Jones D, Textor S, Goff DC, Murphy TP, Toto RD, White A, Cushman WC, White W, Sica D, Ferdinand K, Giles TD, Falkner B, Carey RM; American Heart Association Professional Education Committee. Resistant hypertension: diagnosis, evaluation, and treatment: a scientific statement from the American Heart Association Professional Education Committee of the Council for High Blood Pressure Research. Circulation. 2008 Jun 24;117(25):e510-26. doi: 10.1161/CIRCULATIONAHA.108.189141. PMID 18574054
- [Background] DiBona GF. Sympathetic nervous system and the kidney in hypertension. Curr Opin Nephrol Hypertens. 2002 Mar;11(2):197-200. doi: 10.1097/00041552-200203000-00011. PMID 11856913
- [Background] DiBona GF, Kopp UC. Neural control of renal function. Physiol Rev. 1997 Jan;77(1):75-197. doi: 10.1152/physrev.1997.77.1.75. PMID 9016301
- [Background] Esler M, Jennings G, Korner P, Willett I, Dudley F, Hasking G, Anderson W, Lambert G. Assessment of human sympathetic nervous system activity from measurements of norepinephrine turnover. Hypertension. 1988 Jan;11(1):3-20. doi: 10.1161/01.hyp.11.1.3. No abstract available. PMID 2828236
- [Background] Schlaich MP, Lambert E, Kaye DM, Krozowski Z, Campbell DJ, Lambert G, Hastings J, Aggarwal A, Esler MD. Sympathetic augmentation in hypertension: role of nerve firing, norepinephrine reuptake, and Angiotensin neuromodulation. Hypertension. 2004 Feb;43(2):169-75. doi: 10.1161/01.HYP.0000103160.35395.9E. Epub 2003 Nov 10. PMID 14610101
- [Background] MORRISSEY DM, BROOKES VS, COOKE WT. Sympathectomy in the treatment of hypertension; review of 122 cases. Lancet. 1953 Feb 28;1(6757):403-8. doi: 10.1016/s0140-6736(53)91589-x. No abstract available. PMID 13024041
- [Background] SMITHWICK RH, THOMPSON JE. Splanchnicectomy for essential hypertension; results in 1,266 cases. J Am Med Assoc. 1953 Aug 15;152(16):1501-4. doi: 10.1001/jama.1953.03690160001001. No abstract available. PMID 13061307
- [Background] Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Modification of Diet in Renal Disease Study Group. Ann Intern Med. 1999 Mar 16;130(6):461-70. doi: 10.7326/0003-4819-130-6-199903160-00002. PMID 10075613
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. National Heart, Lung, and Blood Institute; National High Blood Pressure Education Program Coordinating Committee. Seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. Hypertension. 2003 Dec;42(6):1206-52. doi: 10.1161/01.HYP.0000107251.49515.c2. Epub 2003 Dec 1. PMID 14656957
- [Background] Grassi G, Seravalle G, Quarti-Trevano F, Dell'Oro R, Bombelli M, Cuspidi C, Facchetti R, Bolla G, Mancia G. Adrenergic, metabolic, and reflex abnormalities in reverse and extreme dipper hypertensives. Hypertension. 2008 Nov;52(5):925-31. doi: 10.1161/HYPERTENSIONAHA.108.116368. Epub 2008 Sep 8. PMID 18779438
- [Background] DiBona GF. Renal innervation and denervation: lessons from renal transplantation reconsidered. Artif Organs. 1987 Dec;11(6):457-62. doi: 10.1111/j.1525-1594.1987.tb02710.x. PMID 3326559
- [Background] Hausberg M, Kosch M, Harmelink P, Barenbrock M, Hohage H, Kisters K, Dietl KH, Rahn KH. Sympathetic nerve activity in end-stage renal disease. Circulation. 2002 Oct 8;106(15):1974-9. doi: 10.1161/01.cir.0000034043.16664.96. PMID 12370222
- [Background] Schlaich MP, Socratous F, Hennebry S, Eikelis N, Lambert EA, Straznicky N, Esler MD, Lambert GW. Sympathetic activation in chronic renal failure. J Am Soc Nephrol. 2009 May;20(5):933-9. doi: 10.1681/ASN.2008040402. Epub 2008 Sep 17. PMID 18799718
- [Background] DiBona GF. Neural control of the kidney: past, present, and future. Hypertension. 2003 Mar;41(3 Pt 2):621-4. doi: 10.1161/01.HYP.0000047205.52509.8A. Epub 2002 Dec 16. PMID 12623969
- [Background] Fagius J. Sympathetic nerve activity in metabolic control--some basic concepts. Acta Physiol Scand. 2003 Mar;177(3):337-43. doi: 10.1046/j.1365-201X.2003.01086.x. PMID 12609004
- [Background] Joles JA, Koomans HA. Causes and consequences of increased sympathetic activity in renal disease. Hypertension. 2004 Apr;43(4):699-706. doi: 10.1161/01.HYP.0000121881.77212.b1. Epub 2004 Feb 23. PMID 14981063
- [Background] Luippold G, Beilharz M, Muhlbauer B. Chronic renal denervation prevents glomerular hyperfiltration in diabetic rats. Nephrol Dial Transplant. 2004 Feb;19(2):342-7. doi: 10.1093/ndt/gfg584. PMID 14736957
- [Background] Ye S, Zhong H, Yanamadala V, Campese VM. Renal injury caused by intrarenal injection of phenol increases afferent and efferent renal sympathetic nerve activity. Am J Hypertens. 2002 Aug;15(8):717-24. doi: 10.1016/s0895-7061(02)02959-x. PMID 12160195
- [Background] Campese VM, Kogosov E, Koss M. Renal afferent denervation prevents the progression of renal disease in the renal ablation model of chronic renal failure in the rat. Am J Kidney Dis. 1995 Nov;26(5):861-5. doi: 10.1016/0272-6386(95)90456-5. PMID 7485145
- [Background] Prochnau D, Lucas N, Kuehnert H, Figulla HR, Surber R. Catheter-based renal denervation for drug-resistant hypertension by using a standard electrophysiology catheter. EuroIntervention. 2012 Jan;7(9):1077-80. doi: 10.4244/EIJV7I9A171. PMID 21959556
- [Background] Brandt MC, Mahfoud F, Reda S, Schirmer SH, Erdmann E, Bohm M, Hoppe UC. Renal sympathetic denervation reduces left ventricular hypertrophy and improves cardiac function in patients with resistant hypertension. J Am Coll Cardiol. 2012 Mar 6;59(10):901-9. doi: 10.1016/j.jacc.2011.11.034. PMID 22381425
- [Background] EVELYN KA, SINGH MM, CHAPMAN WP, PERERA GA, THALER H. Effect of thoracolumbar sympathectomy on the clinical course of primary (essential) hypertension. A ten-year study of 100 sympathectomized patients compared with individually matched, symptomatically treated control subjects. Am J Med. 1960 Feb;28:188-221. doi: 10.1016/0002-9343(60)90184-4. No abstract available. PMID 13821037

RESULTS

PARTICIPANT FLOW:
Groups:
- Renal Denervation Group: Celcius Thermacool Catheter or Chilli II Cooled Ablation Catheter based on physician preference: Saline-Irrigated Radiofrequency Ablation Catheter placed in the renal arteries in a circumferential manner and energy delivered to create 4 burn lesions.
Period: Overall Study
Arm/Group | Renal Denervation Group
Started | 38
Completed | 20
Not Completed | 18
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 10
Not completed — Screen failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Renal Denervation Group
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Ambulatory Systolic Blood Pressure
Description: The change in systolic blood pressure as measured by 24 hour ambulatory monitoring at 6 months as compared to from baseline.
Time Frame: baseline and 6 months
Population: analysis for participants who returned for follow up
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation Group
Number analyzed (Participants) | 17
mmHg | -10.2 (16.4)

2. Primary Outcome: Change in Ambulatory Diastolic Blood Pressure
Description: The change in diastolic blood pressure as measured by 24 hour ambulatory monitoring at 6 months as compared to from baseline.
Time Frame: baseline and 6 months
Population: analysis for participants who returned for follow up
Measure: Mean (Standard Deviation); unit: mmHg mean change
Arm/Group | Renal Denervation Group
Number analyzed (Participants) | 17
mmHg mean change | -5.5 (9.8)

3. Secondary Outcome: Office Systolic BP
Description: Different time points office systolic blood pressure measurements
Time Frame: baseline, 6 month, 12 months
Population: some participants withdrew from the study, and others were lost to follow up.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Renal Denervation Group
Number analyzed (Participants) | 38
mm Hg
  Baseline | 156.86 (24.3)
  6 months: number analyzed (Participants) | 27
  6 months | 151.19 (28.6)
  12 months: number analyzed (Participants) | 20
  12 months | 158.45 (27.1)

4. Secondary Outcome: Office Diastolic BP
Description: Different time points office diastolic blood pressure measurements
Time Frame: baseline, 6 month, 12 months
Population: some participants withdrew from the study, and others were lost to follow up.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Renal Denervation Group
Number analyzed (Participants) | 38
mm Hg
  Baseline | 87.06 (17.9)
  6 months: number analyzed (Participants) | 27
  6 months | 86.93 (19.3)
  12 months: number analyzed (Participants) | 20
  12 months | 87.75 (14.3)

5. Secondary Outcome: Renal Aortic Ratio
Description: Renal artery blood flow as measured by Renal Aortic Ratio (RAR) = Peak systolic Velocity renal artery / Peak Systolic Velocity Aorta. A >60% stenosis is reported when there is a >3.5:1 Renal to Aortic Ratio.
Time Frame: Baseline and 12 months
Population: Some participants withdrew from the study, others were lost to follow up
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Renal Denervation Group
Number analyzed (Participants) | 28
ratio
  Baseline Right RAR | 1.38 (0.48)
  Baseline Left RAR | 1.52 (0.39)
  12 months Right RAR: number analyzed (Participants) | 15
  12 months Right RAR | 1.41 (0.59)
  12 months Left RAR: number analyzed (Participants) | 15
  12 months Left RAR | 1.52 (0.53)

6. Secondary Outcome: Resistive Index
Description: Renal artery blood flow as measured by Resistive Index. RI = (peak systolic velocity - end diastolic velocity ) / peak systolic velocity. the normal value is ~ 0.60, with 0.70 being around the upper limits of normal
Time Frame: Baseline and 12 months
Population: Some participants withdrew from the study, others were lost to follow up
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Renal Denervation Group
Number analyzed (Participants) | 28
index
  Baseline Right RI | 0.67 (0.16)
  Baseline Left RI | 0.72 (0.12)
  12 months Right RI: number analyzed (Participants) | 15
  12 months Right RI | 0.72 (0.08)
  12 months Left RI | 0.72 (0.09)

7. Secondary Outcome: Renal Artery Dimensions
Description: Dimensions of renal artery, right and left
Time Frame: baseline and 12 months
Population: some participants withdrew from the study, some were lost to follow up
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Renal Denervation Group
Number analyzed (Participants) | 28
mm
  Baseline R Kidney | 11.43 (1.37)
  Baseline L Kidney | 11.68 (1.36)
  12 months R Kidney: number analyzed (Participants) | 15
  12 months R Kidney | 11.26 (1.76)
  12 months L Kidney: number analyzed (Participants) | 15
  12 months L Kidney | 11.39 (1.67)

8. Secondary Outcome: Blood Urea Nitrogen
Description: A blood urea nitrogen (BUN) test measures the amount of nitrogen in blood that comes from the waste product urea. Urea is made when protein is broken down in the body. Urea is made in the liver and passed out in the urine.
Time Frame: baseline, 6 months, 12 months
Population: some participants withdrew from the study, others were lost to followup
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Renal Denervation Group
Number analyzed (Participants) | 38
mg/dL
  Baseline | 20.82 (8.3)
  6 months: number analyzed (Participants) | 26
  6 months | 22.15 (8.49)
  12 months: number analyzed (Participants) | 19
  12 months | 23.11 (15.4)

9. Secondary Outcome: Creatinine
Description: Creatinine measures the level of the waste product in the body. The amount of creatinine in the blood depends partly on the amount of muscle tissue you have. Men generally have higher creatinine levels than women.Normal levels of creatinine in the blood are approximately 0.6 to 1.2 milligrams (mg) per deciliter (dL) in adult males and 0.5 to 1.1 milligrams per deciliter in adult females. High levels of creatinine indicates kidney impairment.
Time Frame: baseline, 6 months, 12 months
Population: some participants withdrew from the study, others were lost to followup
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Renal Denervation Group
Number analyzed (Participants) | 38
mg/dl
  Baseline | 1.6 (1.8)
  6 months: number analyzed (Participants) | 26
  6 months | 1.68 (2.05)
  12 months: number analyzed (Participants) | 19
  12 months | 2.03 (2.8)

10. Secondary Outcome: Anti-hypertensive Medications
Description: The total number of anti-hypertensive medications at baseline, 6 months, and 12 months
Time Frame: Baseline, 6 months, 12 months
Population: some participants withdrew from the study, some were lost to follow-up
Measure: Mean (Standard Deviation); unit: medications
Arm/Group | Renal Denervation Group
Number analyzed (Participants) | 38
medications
  Baseline | 5.37 (1.46)
  6 months: number analyzed (Participants) | 29
  6 months | 4.79 (1.29)
  12 months: number analyzed (Participants) | 22
  12 months | 4.64 (1.6)

ADVERSE EVENTS:
Arm/Group | Renal Denervation Group
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 18/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Renal Denervation Group (N=20)
Elevated Blood Pressure or Hypertensive Crisis (Cardiac disorders) | 8
Atrial Fibrillation (Cardiac disorders) | 3
Penumonia and/or sepsis (Reproductive system and breast disorders) | 3
Renal Artery Dissection (Renal and urinary disorders) | 1
Cerebravascular Accident (Nervous system disorders) | 1
Transient Ischemic Attack (Nervous system disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Renal Denervation Group (N=20)
Diarrhea (Gastrointestinal disorders) | 3
Right Groin Pain (Renal and urinary disorders) | 3
Chest Pain (Cardiac disorders) | 2
Dyspnea (Cardiac disorders) | 2
Syncope (Cardiac disorders) | 2
Groin Hematoma (Renal and urinary disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Bilateral Lower Extremity Edema (Cardiac disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Abdominal Discomfort (Musculoskeletal and connective tissue disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Difficulty Swallowing (Gastrointestinal disorders) | 1
Right Femoral Area Pain (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes